CLINICAL TRIAL: NCT02044666
Title: Pilot Safety Study of Micronized Small Intestinal Submucosa (SIS) for Critical Limb Ischemia
Brief Title: Cook Micronized Small Intestinal Submucosa (SIS) for Critical Limb Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-004
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Ischemia; Peripheral Arterial Disease; Peripheral Vascular Diseases
Keywords: Critical Limb Ischemia; Amputation
MeSH Terms: conditions — Ischemia; Peripheral Arterial Disease; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Micronized Small Intestinal Submucosa (SIS)

INTERVENTIONS:
Device: Micronized Small Intestinal Submucosa (SIS) — Micronized Small Intestinal Submucosa (SIS)

SUMMARY:
This study is intended to collect safety and effectiveness data on the Cook Micronized Small Intestinal Submucosa (SIS)

ELIGIBILITY:
Inclusion Criteria:

* Rutherford stage 4 or 5 or Leriche-Fontaine classification IIIB
* Patient is unable to be treated by endovascular or surgical means

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient has had a previous surgery within 30 days of the study procedure
* Patient has a planned surgical or interventional procedure within 30 days after the study procedure
* Patient has a life expectancy of less than 1 year
* Patient has a known allergy to pigs or pig products, or has a religious or cultural objection to the use of pig tissue.
* Additional restrictions as specified in the protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Frequency and types of adverse events | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Kong Teng Tan, MD, Principal Investigator — Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada